CLINICAL TRIAL: NCT00877331
Title: Brief Intervention in Primary Care for Problem Drug Use and Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Peter Roy-Byrne, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34892-C; R01DA026014 (NIH)
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Substance-Related Disorders
Keywords: Drug Abuse; Drug Addiction; Drug Dependence; Drug Usage; Drug Use Disorders; Substance Abuse; Substance Addiction; Substance Dependence; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Brief intervention using motivational interviewing. One in-person session (30-45 minutes) with a brief phone follow-up one week later.
  Interventions: Behavioral: Brief intervention using motivational interviewing
- 2 (No Intervention): Enhanced care as usual.

INTERVENTIONS:
Behavioral: Brief intervention using motivational interviewing — One brief, in-person motivational interviewing session (30-45 minutes) in conjunction with the medical appointment. Plus one brief follow-up phone call one week later.
  Arms: 1

SUMMARY:
This study will examine the effectiveness of a brief intervention in a primary care setting to reduce drug use or abuse compared to enhanced care as usual.

DETAILED DESCRIPTION:
A substantial body of research has established the efficacy and effectiveness of brief interventions (BI) for excessive or "hazardous" alcohol use in patients seen in medical settings. Dissemination projects of brief interventions for alcohol and drugs have recently been implemented on a widespread scale. This rapid progression of brief intervention for drugs other than alcohol has outstripped its evidence base.

The aims of the study as outlined in the grant are:

1. To examine whether BI is effective at improving outcomes (self-reported drug use and attendance in drug abuse treatment) in individuals with a wide range of problem drug use over and above enhanced care as usual. The enhanced control condition will consist of routine screening, patient notification, and referral for treatment.
2. To test whether fidelity to the BI model or lower severity of drug use is associated with better outcomes.
3. To estimate the impact of BI on several public health outcomes that are directly related to the hazardous effects of illicit drug use, including the use of acute health care services, involvement in the criminal justice system, employment, HIV risk behavior, and mortality.
4. To estimate the costs of the intervention, potential cost offsets, and its incremental cost-effectiveness versus enhanced usual care from the payer perspective based on health care service use and drug use frequency.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* receive medical care at one of the participating primary care clinics at Harborview Medical Center/University of Washington Medical Center
* will maintain care at the clinic for one year
* have a phone or easy access to phone, voicemail, or email
* used recreational drugs in the last 3 months
* used prescription medications not as prescribed in the last 3 months

Exclusion Criteria:

* participation in any formal substance abuse treatment programs in the last 30 days (excluding 12-step or self-help groups)
* terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2009-04; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Use of illicit drugs in the past 30 days | baseline, 3, 6, 9, and 12 months
  Use of illicit drugs in the past 30 days will be measured by self-reported days of use in the past 30 days and validated by urine toxicological screen.
Enrollment in formal substance abuse treatment | baseline up to 2 years post-intervention
  Enrollment in formal substance abuse treatment will be measured as an admission to chemical dependency treatment as recorded in the Washington State TARGET database.
Medical, legal, employment, social, and psychiatric outcomes | baseline, 3, 6, 9, and 12 months
  Medical, legal, employment, social, and psychiatric outcomes will be measured by composite scores on the Addiction Severity Index (ASI) Lite.

SECONDARY OUTCOMES:
Public health outcomes | baseline up to 2 years post-intervention
  Public health outcomes will be measured by administrative data sources (emergency room visits, hospitalizations, hospital days, HIV risk behavior, arrests, and death).
Cost of the intervention | baseline up to 2 years post-intervention
  Cost of the intervention will be measured using methods previously employed in the COMBINE study.
Incremental cost-effectiveness | baseline up to 2 years post-intervention
  Incremental cost-effectiveness will be measured from the payer perspective based on health care service use and drug use frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Roy-Byrne, MD, Principal Investigator — University of Washington; Kristin Bumgardner, BS, Study Director — University of Washington; Antoinette Krupski, PhD, Study Chair — University of Washington; Richard Ries, MD, Study Chair — University of Washington; Chris Dunn, PhD, Study Chair — University of Washington; Dennis Donovan, PhD, Study Chair — University of Washington; Jutta M. Joesch, PhD, Study Chair — University of Washington; Gary A. Zarkin, PhD, Study Chair — RTI International
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Krupski A, Joesch JM, Dunn C, Donovan D, Bumgardner K, Lord SP, Ries R, Roy-Byrne P. Testing the effects of brief intervention in primary care for problem drug use in a randomized controlled trial: rationale, design, and methods. Addict Sci Clin Pract. 2012 Dec 14;7(1):27. doi: 10.1186/1940-0640-7-27. PMID 23237456
- [Result] Roy-Byrne P, Bumgardner K, Krupski A, Dunn C, Ries R, Donovan D, West II, Maynard C, Atkins DC, Graves MC, Joesch JM, Zarkin GA. Brief intervention for problem drug use in safety-net primary care settings: a randomized clinical trial. JAMA. 2014 Aug 6;312(5):492-501. doi: 10.1001/jama.2014.7860. PMID 25096689